CLINICAL TRIAL: NCT04456829
Title: Investigation of the Efficacies of a Resveratrol Formula on Improvement of Skin
Brief Title: Investigation of the Efficacies of a Resveratrol Formula on Improvement of Skin Conditions and Inflammatory Related Factors
Acronym: Resveratrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-0-54-B
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Skin Conditions; Proinflammatory Cytokines
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol drink (Experimental)
  Interventions: Dietary Supplement: Resveratrol drink
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Resveratrol drink — Subjects will consume a bottle of resveratrol drink for two months.
  Other Names: Grape Yeast Compound Fruit Vegetable Beverage
  Arms: Resveratrol drink
Dietary Supplement: Placebo drink — Subjects will consume a bottle of placebo drink for two months.
  Arms: Placebo drink

SUMMARY:
To assess a resveratrol formula on improvement of skin conditions and inflammatory cytokines in blood

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, heart, liver, kidney, endocrine and other organs and patients with mental illness (according to medical history).
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure in the past 4 weeks.
* Subjects who have large spots (area >3 square centimeter) or abnormal acne.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The change of skin moisture | 0, 4, and 8 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin elasticity | 0, 4, and 8 weeks
  Cutometer® dual MPA 580 was utilized to measure skin elasticity (parameter R2). Units: μm penetration depth into the probe opening, expressed as curves
The change of skin wrinkles | 0, 4, and 8 weeks
  VISIA Complexion Analysis System was utilized to measure wrinkles. Units: arbitrary units
The change of skin collagen density | 0, 4, and 8 weeks
  DermaLab® USB - 20 MHz High Freq. Ultrasound probe was utilized to scan and analyze skin collagen density. Units:
  Intensity score
The change of skin texture | 0, 4, and 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin pores | 0, 4, and 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin pores. Units: arbitrary units
The change of total antioxidant capacity of blood | 0 and 8 weeks
  Total Antioxidant Capacity Assay Kit
The change of TNF-alpha of blood | 0 and 8 weeks
  ELISA Kit
The change of IL-6 of blood | 0 and 8 weeks
  ELISA Kit
The change of IL-17 of blood | 0 and 8 weeks
  ELISA Kit
The change of IL-1β of blood | 0 and 8 weeks
  ELISA Kit

CONTACTS AND LOCATIONS:
Locations (1):
- Chia Nan University of Pharmacy & Science, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No